CLINICAL TRIAL: NCT06555367
Title: Clinical Application Research of Scleral Lenses in Ocular Surface Diseases
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0667
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Ocular Surface Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scleral lenses group: The case group consists of patients with irregular corneas who wear scleral lenses.
  Interventions: Device: scleral lenses
- control group: The control group comprises patients with irregular corneas who have not undergone treatment with scleral lenses.

INTERVENTIONS:
Device: scleral lenses — Wear scleral lenses
  Groups: scleral lenses group

SUMMARY:
To evaluate the therapeutic efficacy of scleral lenses in patients with irregular corneal astigmatism stemming from ocular surface diseases (OSD), focusing on visual acuity improvement, comfort, and overall satisfaction. This prospective clinical study enrolled patients diagnosed with OSD-related irregular corneal astigmatism. Participants underwent comprehensive ophthalmic evaluation, including corneal topography, visual acuity assessment, and tear film analysis. Qualified subjects were fitted with scleral lenses and followed up at intervals of one week, one month, and three months post-fitting. The primary outcomes measured were uncorrected and corrected visual acuity, comfort levels assessed via a standardized questionnaire, and fitting success rates. Data were analyzed using appropriate statistical methods to compare pre- and post-intervention values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with irregular corneal astigmatism, including those with post-keratoconus cross-linking surgery, post-keratoplasty, and corneal irregularities caused by trauma; Volunteers who are willing to participate in this trial, have signed the informed consent form, and are willing to cooperate with the treatment and follow-up; Individuals aged 18 years or older (including 18 years old), with no gender restrictions; Cases collected from January 2023 to August 2024.

Exclusion Criteria:

* Unable or unwilling to sign the consent form, or unable to follow the study procedures; Nursing or pregnant women; Individuals with acute ocular inflammation or infection; Corneal endothelium: Cell Density (CD) <1000/mm²; Individuals required to wear lenses overnight; Poor compliance; Those who do not meet the hygiene requirements for lens wear; Individuals whom the investigator deems have other reasons making them unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with irregular corneal astigmatism who visited the ophthalmology clinic of the Second Affiliated Hospital of Zhejiang University for scleral lens fitting from January 2022 to June 2024 were selected. This includes patients with post-keratoconus cross-linking surgery, post-keratoplasty, and those with corneal irregularities caused by trauma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-08 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Scleral lens fitting assessment | 4 hours later
  The fitting assessment is conducted using a slit lamp microscope to observe the central positioning of the lens, the tear film space under the lens, and the vascular compression on the peripheral conjunctival surface. OCT is applied to measure the tear film space between the central and peripheral non-contact areas of the lens and the anterior corneal surface, as well as the landing zone of the lens in all peripheral directions.

SECONDARY OUTCOMES:
Subjective comfort assessment | 4 hours later
  Level 1: Very uncomfortable; Level 2: Uncomfortable; Level 3: Moderate comfort; Level 4: Comfortable; Level 5: Very comfortable.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University Hospital, Hangzhou, Zhejiang, China